CLINICAL TRIAL: NCT02538068
Title: Meaning and Purpose as Predictors of Physical Activity Maintenance
Brief Title: The Psychology of Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-0275; 14PRE18710033 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2015-08-21; First posted 2015-09-02 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Sedentary Lifestyle
Keywords: Purpose in Life; Self-determination; Physical activity; Self-monitoring; Behavior change
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily Surveys (Experimental): Participants complete a daily survey regarding their daily life meaning, mood, physical activity, and other activities for 4 weeks.
  Interventions: Behavioral: Daily Surveys
- Random Surveys (8) (Active Comparator): Participants complete 8 random surveys over the first 4 weeks.
  Interventions: Behavioral: Random Surveys (8)

INTERVENTIONS:
Behavioral: Daily Surveys — Participants complete 28 daily surveys of daily meaning, mood, and physical activities.
  Arms: Daily Surveys
Behavioral: Random Surveys (8) — Participants complete 8 random surveys of activities over the past 24 hours during the first 4 weeks.
  Arms: Random Surveys (8)

SUMMARY:
This study plans to learn more about psychosocial factors that contribute to adopting physical activity. The goal of this study is to improve upon existing theories of behavior change in order to help other people become more physically active.

DETAILED DESCRIPTION:
The purpose of this study is to examine the relationship between personal life meaning and purpose and physical activity maintenance in a group of previously sedentary adults starting new exercise programs. Participants complete questionnaires at baseline, 4 weeks, and 12 weeks after starting an exercise program. Participants are randomly assigned to complete questionnaires about daily meaning, mood, and activity for the first 4 weeks or to complete 8 random questionnaires about daily activities over the first 4 weeks. It is hypothesized that personal life meaning and purpose will be related to greater exercise participation at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 30-89 years old
* Joining or already a member of the Anschutz Health and Wellness Fitness Center
* Able to read and understand English
* Sedentary (< 60 minutes of moderate-vigorous physical activity a week) for the past 3 months
* Planning to start a new exercise program

Exclusion Criteria:

* Physical contraindications to participate in physical activity (as defined as a positive PAR-Q score)
* Existing diagnosis of cardiovascular disease
* Currently pregnant

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in Physical Activity as measured by the International Physical Activity Questionnaire - Short Form | Baseline, 4 weeks, and 12 weeks
  Evaluation of Physical Activity as measured by the International Physical Activity Questionnaire - Short Form

SECONDARY OUTCOMES:
Frequency of Fitness Center Attendance measured by number of check-ins at fitness center | Daily for 12 weeks
  Number of check-ins at fitness center over 12 weeks
Changes in Physical Fitness, as measured by a combined scores on objective cardiovascular fitness, flexibility, and strength. | Baseline and 12 weeks
  Evaluate changes in cardiovascular, flexibility and strength. Participants complete a YMCA 3-minute step test for cardiovascular fitness (assessment of resting heart rate and recovery heart rate), a sit-and-reach test for flexibility, and a grip strength test for strength. Participants objective scores on these tests will be categorized on scales from 1 (poor fitness) to 5 (excellent fitness) based on age and gender and combined for a total fitness score (ranging from 4 to 20).

OTHER OUTCOMES:
Changes in the Satisfaction with Life assessed by Satisfaction of Life Scale | Baseline, 4 weeks, and 12 weeks
  The subject's satisfaction with life will be assessed by completing a Satisfaction of Life Scale.
Changes in Vitality assessed by Subjective Vitality Scale | Baseline, 4 weeks, and 12 weeks
  Vitality will be assessed by completing a Subjective Vitality Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Hooker, MS, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Derived] Hooker SA, Masters KS. Daily meaning salience and physical activity in previously inactive exercise initiates. Health Psychol. 2018 Apr;37(4):344-354. doi: 10.1037/hea0000599. Epub 2018 Jan 25. PMID 29369678